CLINICAL TRIAL: NCT04781205
Title: Operating Community Primary Care Clinics Under Personalized Medicine Paradigm and Determining Differences in Health Outcomes Between Clinics With and Without Intervention.
Brief Title: Genome Driven Primary Care Clinics - an RCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Gad Rennert, Professor and Chairman, Dept. of Community Medicine and Epidemiology, Carmel Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CMC-16-0071-CTIL
Record Dates: First submitted 2021-02-14; First posted 2021-03-04 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-02

CONDITIONS: Health Services Administration; Genetic Predisposition; Microbial Colonization
Keywords: wearable monitors, microbiome, genomic medicine,
MeSH Terms: conditions — Genetic Predisposition to Disease; Communicable Diseases | interventions — Genome-Wide Association Study; Whole Genome Sequencing

STUDY DESIGN:
Intervention Model Description: Paired cluster randomization of 40 clinics into 20 intervention and 20 usual care. Randomization from among a couple of similar clinics
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Members of clinics randomized into intervention arm will be consented on a blood test for DNA evaluation (up to WGS), a single feces sample for microbiome analysis and tentative agreement to ware monitors of various vital signs of body function
  Interventions: Genetic: Mutation arrays, NGS panels, GWAS, WES, WGS,; Device: wearable monitors
- Usual care (No Intervention): No intervention at all

INTERVENTIONS:
Genetic: Mutation arrays, NGS panels, GWAS, WES, WGS, — DNA extracted from peripheral blood as well as genetic analysis of bacteria from feces
  Arms: Intervention
Device: wearable monitors — test various technologies of sensors to measure continuously various body functions and provide information to person and to physician
  Arms: Intervention

SUMMARY:
A cluster randomized controlled study of 40 primary care clinics in Northern Israel (20 intervention clinics, 20 usual care clinics) to evaluate the value of introducing a precision medicine/genomic approach/paradigm on the clinical and economical outcomes of the clinics. Intervention includes 3 elements: 1. DNA extraction and evaluation (up to the level of WGS); 2. Feces sample for microbiome study, 3. Wearable devices for continuous monitoring of body functions. Expected number of participants is 100,000 in each arm. Results will be calculated for a clinic as a unit and not for individuals (each clinic to be compared to "twin" selected clinic).

DETAILED DESCRIPTION:
Study major aim:

Assess whether employing a paradigm of genomic/precision medicine in primary care clinics can lead to an improvement in the medical or economic outcomes of the clinic as a unit.

Specific and secondary aims

1. Study differences in morbidity, mortality, quality of life or the cost of medical service indicators between clinics operating under a genome driven paradigm compared to usual care clinics.
2. Examine whether the public has an interest in extensive genetic testing.
3. Examine whether the medical staff has an interest and ability to assimilate a genomic approach in the routine clinic work.
4. Identify links between genetic markers (mutations, variants) and different diseases (incidence or clinical behavior) or different drug responses (resistance, effectiveness, side-effects).
5. Examine whether the implementation of prolonged personal monitoring devices will lead to improved morbidity and mortality indices.
6. Examine whether measuring genomic variability in the microbiome has implications on health status or means of coping with different diseases and different health conditions.

ELIGIBILITY:
Inclusion Criteria:

* All clinic adult population
* All diseases

Exclusion Criteria:

* Mentality unable to understand and sign consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200000 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
chronic diseases in clinic | 5 years
  whole clinic Incidence rate/100,000 of major chronic diseases (hypertension, Hyperlipidemia, DM, IHD, Cancer)
Mortality in clinic | 5 ytears
  whole clinic mortality rate/100,000 of major chronic diseases (DM, cancer, IHD)
costs in clinic | 5 years
  Total annual cost of clinic activity in NIS, including cost of diagnostic tests and hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Gad Rennert, MD, PhD, Principal Investigator — Clalit National Cancer Control Center Carmel Medical Center, Technion,
Locations (1):
- Carmel Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No
study comparative unit is a whole clinic and not an individual participants